CLINICAL TRIAL: NCT00628888
Title: Treatment of Emotional Disorders in Adolescence
Brief Title: A Waitlist-Controlled Trial of the Unified Protocol for the Treatment of Emotional Disorders in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jill May Ehrenreich, Associate Professor of Psychology, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K23MH073946 (NIH); K23MH073946 (NIH); DDTR BK-TKPD
Record Dates: First submitted 2008-02-29; First posted 2008-03-05 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Anxiety Disorders; Depression
Keywords: Unipolar Depression; Anxiety; Adolescent; Emotion; Cognitive Behavioral
MeSH Terms: conditions — Anxiety Disorders; Depression; Depressive Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Unified Protocol for Adolescents (UP-A) (Experimental): Participants receive the UP-A intervention for 8-21 weeks immediately following randomization.
  Interventions: Behavioral: Unified Protocol for Adolescents (UP-A)
- Delayed Treatment/Waitlist (Experimental): Participants receive an 8-week waitlist condition with some attentional-control via monitoring for clinical deterioration. After a post-waitlist assessment, participants in this condition are offered the UP-A treatment for 8-21 weeks.
  Interventions: Behavioral: Unified Protocol for Adolescents (UP-A)

INTERVENTIONS:
Behavioral: Unified Protocol for Adolescents (UP-A) — All participants will be offered the UP-A intervention, inclusive of 8 and 21 weekly sessions of an emotion-focused treatment with cognitive-behavioral elements, either immediately following randomization or after an 8-week delayed treatment waitlist. The UP-A sessions are delivered in a flexible manner. Several of the UP-A's treatment elements are fixed and received by all participants (psychoeducation about emotions and emotional behavior, awareness and mindfulness skills, antecedent cognitive reappraisal/problem-solving skills, emotion exposure strategies, and relapse prevention skills), although applied for varying numbers of sessions depending on clinical need. Other strategies (motivational enhancement, parenting strategies and crisis management strategies) are applied on an as-needed basis based on client needs.
  Other Names: Emotion Regulation; Evidence Based Treatment

SUMMARY:
This study will evaluate the effectiveness of an emotion-focused cognitive behavioral treatment program for adolescents with anxiety or unipolar depressive disorders.

DETAILED DESCRIPTION:
Anxiety and depression are among the most prevalent psychiatric disorders in youth. Adolescents with anxiety or depression experience persistent emotional distress that can cause problems with school, family, and friends. In addition, anxiety and depressive disorders commonly co-exist, causing further distress for those affected. If left untreated, the difficulties associated with these disorders can persist into adulthood. Fortunately, anxiety and depression are highly treatable using a combination of medications and forms of psychotherapy, but many youth in community settings are unlikely to receive these treatments. An emotion-focused, cognitive behavioral treatment, specifically designed to meet a broad range of treatment needs of adolescents, may provide one way of translating effective treatment components to community settings. This study will evaluate the effectiveness of a transdiagnostic, emotion-focused, cognitive behavioral treatment program, called the Unified Protocol for the Treatment of Emotional Disorders in Adolescents (UP-A), for youth with anxiety or unipolar depressive disorders.

Participants in this study will be assigned to receive either immediate or delayed UP-A program sessions. Study participation will last up to 12 months after beginning treatment. Upon initiation of treatment, parent and child participants will undergo initial assessments that will include questionnaires about anxiety, worry, depression and emotion regulation; and an interview pertaining to the adolescent's anxiety and depression. Both parent and adolescent participants will then attend up to 21 weekly treatment sessions, lasting 60 minutes each. During sessions, participants will learn skills regarding acceptance of intense emotional states, how to actively cope with emotions, and act in healthy ways during anxiety- and depression-provoking situations. Throughout the course of treatment, parent and adolescent participants will be asked to keep records about the adolescent's emotions and functioning. Participants will also be given at-home assignments to practice skills learned in treatment sessions. During and after treatment, participants will complete questionnaires about their thoughts on the treatment sessions. Participants will repeat the initial assessment either following the waitlist delayed treatment condition or 8 weeks into treatment, immediately after the last treatment session as well as at months 3 and 6 of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Principal diagnosis of major depressive disorder, social anxiety disorder, social phobia, panic disorder with or without agoraphobia, generalized anxiety disorder, obsessive compulsive disorder, agoraphobia, post-traumatic stress disorder, dysthymic disorder, anxiety disorder not-otherwise-specified, or depressive disorder not-otherwise-specified
* At least one parent (or caregiver with whom the adolescent is living) available to accompany the adolescent to all assessment sessions and attend parent sessions as prescribed
* For adolescents on medication, there must be a 1-month stabilization period (for benzodiazepines) or 3-month stabilization period (for selective serotonin reuptake inhibitors, serotonin-norepinephrine reuptake inhibitors, or tricyclics) before study entry
* Able to maintain current medication regimen (or remain off psychopharmacologic treatment if not currently taking such medications) throughout the study, unless changes are medically necessary

Exclusion Criteria:

* Co-occurring conditions, including positive diagnosis of schizophrenia, bipolar I or II disorder, pervasive developmental disorder, organic brain syndrome, mental retardation , or current suicidal/homicidal ideation
* A prior course of cognitive behavioral treatment
* Inability to speak, read, or understand English sufficiently well to complete study procedures

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2006-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Clinical Severity Rating (CSR) on the Anxiety Disorders Interview Schedule for DSM-IV, child and parent versions (ADIS-IV-C/P) | Measured pre- and post-treatment, post-waitlist or 8 weeks into treatment and 3 and 6 months following treatment
Treatment gains and overall patient functioning measured by: Clinical Global Impression Scale(CGI) | Measured at all post-treatment, waitlist and other follow-up points

SECONDARY OUTCOMES:
Emotion Regulation indices | Measured pre- and post-treatment, post waitlist or 8 weeks into treatment and 3 months and 6 months after treatment
Changes in Anxiety and Depressive symptomology assessed by the CBCL and RCADS (parent and child version) | Measured pre- and post-treatment, post waitlist or 8 weeks into treatment, 3 and 6 months following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jill Ehrenreich-May, PhD, Principal Investigator — University of Miami
Locations (1):
- Child and Adolescent Mood and Anxiety Treatment (CAMAT) Program, Miami, Florida, United States

REFERENCES:
- [Background] Levin L, Henderson HA, Ehrenreich-May J. Interpersonal predictors of early therapeutic alliance in a transdiagnostic cognitive-behavioral treatment for adolescents with anxiety and depression. Psychotherapy (Chic). 2012 Jun;49(2):218-230. doi: 10.1037/a0028265. PMID 22642525
- [Background] Girio-Herrera E, Ehrenreich-May J. Using flexible clinical processes in the Unified Protocol for the Treatment of Emotional Disorders in Adolescence. Psychotherapy (Chic). 2014 Mar;51(1):117-22. doi: 10.1037/a0032517. PMID 24635001
- [Result] Queen AH, Barlow DH, Ehrenreich-May J. The trajectories of adolescent anxiety and depressive symptoms over the course of a transdiagnostic treatment. J Anxiety Disord. 2014 Aug;28(6):511-21. doi: 10.1016/j.janxdis.2014.05.007. Epub 2014 Jun 2. PMID 24960439
- See also: Click here for more information on Dr. Ehnrenreich at the University of Miami Web site — http://www.miami.edu/childanxiety
- See also: Click here for more information on the Child and Adolescent Mood and Anxiety Treatment (CAMAT) program in the Department of Psychology at the University of Miami — http://www.miami.edu/childanxiety